CLINICAL TRIAL: NCT03934177
Title: Impact of Blueberry Consumption on Intestinal Permeability, Gut Microbiota, and Gut-Derived Inflammation in Individuals With Elevated Risk of a Pro-Inflammatory Gut Milieu
Brief Title: Impact of Blueberry Consumption on Gastrointestinal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: Rush University Medical Center (Other); University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 18557
Record Dates: First submitted 2019-04-15; First posted 2019-05-01 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Circadian Dysregulation
Keywords: Blueberry; Microbiota; Intestinal permeability
MeSH Terms: conditions — Obesity; Chronobiology Disorders

STUDY DESIGN:
Intervention Model Description: This 14-week crossover study includes 4 weeks for each of the two supplementation periods (blueberries and placebo), with a 4-week wash out between.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and statistician will blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry powder (Experimental): 4 weeks of supplementation of 24 g whole blueberry powder
  Interventions: Dietary Supplement: Blueberry powder
- Placebo powder (Placebo Comparator): 4 weeks of supplementation of 24 g placebo powder (maltodextrin)
  Interventions: Dietary Supplement: Placebo powder

INTERVENTIONS:
Dietary Supplement: Blueberry powder — Dried, powdered blueberries will be consumed at 24 g/day in two divided doses at least 4 hours apart.
  Arms: Blueberry powder
Dietary Supplement: Placebo powder — A placebo consisting maltodextrin will be consumed at 24 g/day in two divided doses at least 4 hours apart.
  Arms: Placebo powder

SUMMARY:
This study will evaluate the impact of blueberry consumption on markers of gastrointestinal health including gut microbiota, intestinal permeability, and gut-derived inflammation in those vulnerable to a unhealthy gut milieu. All participants will consume a blueberry powder and a placebo in this crossover study.

DETAILED DESCRIPTION:
The commensal bacteria that reside in the human gut, known as the gut microbiota, is a complex system that modulates local gut homeostasis and systemic biological processes. Several environmental factors have been shown to influence the gut milieu (including microbiota), and thus both gastrointestinal and host health. Relevant to the current proposal is the influence of body weight, diet, and circadian rhythms. In the current study, the investigators propose to use these common disruptors of gastrointestinal health through recruiting obese shift workers with a low-fiber diet to identify if these disrupted individuals can benefit from blueberry intake. Specifically, the study objectives are to determine if 24 g whole blueberry powder consumed daily can beneficially modify intestinal permeability, gut microbiota, microbial metabolites, and both gut-derived and systemic inflammation in those most susceptible to a pro-inflammatory milieu. This will be accomplished through a 14-week crossover study in which 28 individuals will be randomized by treatment group order to 4 weeks of whole blueberry powder and placebo powder, with a 4-week wash out in between the treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* obese (BMI +/- 30.0 kg/m2)
* shift workers (shift work overnight (third shift) +/= 3 days/week for the past 3 months)
* 19-70 years of age

Exclusion Criteria:

* patient history of gastrointestinal diseases except for hiatal hernia, GERD, or hemorrhoids, mild gastrointestinal symptoms
* elevated laboratory values from a comprehensive metabolic panel (CMP) and complete blood count (CBC) with the exception of glucose (+/= 126 mg/dL; if elevated, confirmed with HA1c of greater than or equal to 6.5%) and ALT, AST, or ALP over 2 times normal levels (to allow for mild elevations resulting from fatty liver often seen in obese) unless approved by study physician
* currently pregnant or plans to become pregnant during the study as determined by participant report
* antibiotic use within the last 12 weeks prior to enrollment
* presence of chronic metabolic disease (e.g., cardiovascular disease, diabetes, cancer) or per physician discretion
* recent (past 4 weeks) major change in dietary habits or a plan to have a major change in dietary habits during the study
* habitual blueberry consumption of more than 0.5 cups 2x/week or a 4-week washout period if consumes
* allergy or intolerance to blueberries
* consumption of supplemental fiber, probiotics or prebiotics without an appropriate 4-week washout period
* restrictive dietary patterns (e.g., ketogenic, Paleolithic) or a diet high in fiber (+/= 14 g/1000 kilocalories) to increase study result generalizability to the U.S. population (low-fiber diet), as well as provide another stimuli for gut leakiness
* unwillingness to consent to the study.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
intestinal permeability | 28 days
  urinary sugar measurement by gas chromatography (GC): Sucralose, lactulose, mannitol, sucrose as a percent of oral dose.

SECONDARY OUTCOMES:
Microbiota | 28 days
  Microbiota composition through shotgun sequencing. Composition includes relative abundance of all microbes in stool.
Microbial metabolites | 28 days
  Quantity of stool short-chain fatty acid (butyrate, propionate, acetate) per dry stool weight by gas chromatography
Gut-derived/systemic inflammation | 28 days
  Concentration of serum lipopolysaccharide (LPS), LPS-binding protein (LBP), and interleukin-6 (IL6)

CONTACTS AND LOCATIONS:
Overall Officials: Heather E Rasmussen, PhD, Principal Investigator — University of Nebraska Lincoln
Locations (2):
- United States (2):
  - University of Nebraska, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No